CLINICAL TRIAL: NCT00745771
Title: Multiple Dose, Double-Blind, Double-Dummy, Placebo and Active Controlled Study of Pharmacokinetics of Diractin® as Well as Safety and Efficacy for the Treatment of Muscle Soreness From Exercise
Brief Title: Multiple Dose, Double-Blind, Placebo and Active Controlled Study of Pharmacokinetics of Diractin® as Well as Safety and Efficacy for the Treatment of Muscle Soreness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IDEA AG (Industry)
Responsible Party: Ingrid Patzak, IDEA AG
Purpose: Treatment
Other Study IDs: CL-033-II-02
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Muscle Soreness
Keywords: pharmacokinetics; of Diractin®; safety; efficacy; exercise
MeSH Terms: conditions — Myalgia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 200 mg Ketoprofen
  Interventions: Drug: Diractin
- 2 (Active Comparator): 100 mg Ketoprofen
  Interventions: Drug: Diractin

INTERVENTIONS:
Drug: Diractin
  Arms: 1
Drug: Diractin
  Arms: 2

SUMMARY:
Multiple-dose, double-blind, double-dummy, parallel, randomized, placebo and active controlled study of pharmacokinetics of Diractin® as well as safety and efficacy for muscle soreness from exercise.

ELIGIBILITY:
Inclusion Criteria:

* Understands nature and provision of the study

  * Have been informed about the study by the investigator and gave signed and dated informed consent prior to participation
  * Muscle soreness with a pain score of at least 3 on a 10 point categorical pain scale at 12-16h after exercise
  * Male and female subjects
  * Age 18-55 years
  * Subjects in good health as determined by the Investigator
  * Woman of childbearing potential using reliable methods of contraception with a low failure rate (i.e. less than 1% per year), e.g. implants, injectables, combined oral contraceptives, reliable intrauterine-devices, vasectomised/ infertile partner or surgically sterile (uterus removed or both tubes tied) or postmenopausal (at least 2 years without periods)

Exclusion Criteria:

* 4.2.1 General Exclusion Criteria

  * Investigator or any other team member involved directly or indirectly in the conduct of the clinical trial
  * Subjects who are inmates of psychiatric wards, prisons, or other state institutions
  * Participation in another clinical trial within the last 30 days and during the study
  * Not willing to refrain from exposing target areas after treatment to excessive ultraviolet light (solar radiation or solarium)
  * Pregnancy or lactation

4.2.2 Medical History Related Exclusion Criteria

* History of dermal allergic reactions
* Known hypersensitivity or allergy (including photoallergy) to NSAID´s including ketoprofen, and ingredients used in pharmaceutical products
* Alcohol or drug abuse
* Malignancy within the past 2 years
* Skin lesions, dermatological diseases or tattoo in the treatment area
* Major surgery 3 months before enrolment
* NSAID idiosyncrasy
* Impaired haematopoesis and coagulation
* Gastric and duodenal ulcer and gastrointestinal bleedings
* Systemic lupus erythematodes, mixed connective tissue disease
* Major heart disease / uncontrolled hypertension
* Hepatic failure with ALT and/or AST > 2.0 ULN
* Renal failure with serum creatinine levels > 1.5 milligrams/deciliter (mg/dL)
* Varicosis, thrombophlebitis and other vascular disorders of the lower extremities
* Major traumatic lesions (e.g. fracture, tendon or muscle ruptures) of the musculo-sceletal system of the lower limbs
* HIV - Infection
* Hepatitis B or C
* Asthma bronchiale
* Blood donation one month before screening and during study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egbert Seidel, MD, Principal Investigator — X-pert Med Jena
Locations (1):
- X-pert Med GmbH, Jena, Thuringia, Germany